CLINICAL TRIAL: NCT00981032
Title: Improving Implementation of the US Preventive Service Task Force Recommendation for Prophylactic Aspirin Use Among Adults at Risk for Cardiovascular Disease
Brief Title: Improving Aspirin Use Among Adults at Risk for Cardiovascular Disease (CVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Nirav R. Shah, MD, MPH, Geisinger Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-0264
Record Dates: First submitted 2009-09-11; First posted 2009-09-22 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Cardiovascular Disease
Keywords: Aspirin; Behavior; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-visit Summary (Experimental): Patients in this arm will receive a pre-visit summary prior to their appointment. The pre-visit summary details the patient's risk of heart attack or stroke and the benefits of daily prophylactic aspirin use.
  Interventions: Behavioral: Pre-visit Summary
- Clinical Decision Sharing Tool (Experimental): Patients in this arm will receive a pre-visit summary prior to their appointment. They will also view a clinical decision sharing tool in conjunction with the physician in the office. The pre-visit summary details the patient's risk of heart attack or stroke and the benefits of daily prophylactic aspirin use. The clinical decision sharing tool informs the physician of the patient's heart attack or stroke risk and determines if the patient would benefit from aspirin use.
  Interventions: Behavioral: Clinical Decision Sharing Tool

INTERVENTIONS:
Behavioral: Pre-visit Summary — The intervention is a pre-visit summary given to the patient prior to their appointment. The pre-visit summary details the patient's risk of heart attack or stroke and the benefits of daily prophylactic aspirin use.
  Arms: Pre-visit Summary
Behavioral: Clinical Decision Sharing Tool — This intervention includes a pre-visit summary and a clinical decision sharing tool. Patients will receive a pre-visit summary prior to their appointment. They will also view a clinical decision sharing tool in conjunction with the physician in the office. The pre-visit summary details the patient's risk of heart attack or stroke and the benefits of daily prophylactic aspirin use. The clinical decision sharing tool informs the physician of the patient's heart attack or stroke risk and determines if the patient would benefit from aspirin use.
  Arms: Clinical Decision Sharing Tool

SUMMARY:
The investigators' aim is to implement an intervention to increase aspirin prophylaxis use among patients that is patient initiated, optimizes use of physician and staff time, appropriately compensates staff, provides clinicians with tools necessary for managing aspiring prophylaxis, and ensures continuous management.

DETAILED DESCRIPTION:
This intervention addresses a fundamental question of how clinicians need to be directly involved in motivating behavior change (i.e., aspirin prophylaxis). While complex behavior change likely demands high levels of involvement, a single simple action (aspirin prophylaxis) may not require such complex interactions.

We propose to compare the effectiveness of three models of care in a rigorous randomized controlled trial that will consist of a 3-arm, within-clinic design in which patients will be randomized to either the physician-initiated, the patient-initiated model, or to a control group in which usual care is delivered. In a patient-initiated model, patients are active participants in their own care and receive a pre-visit summary that contains an individualized risk assessment and patient education. In the physician-initiated model, patients receive the pre-visit summary and the physician uses a clinical decision support tool through the electronic health record that details the patient risk of CVD.

The specific aims of the proposed work are to compare the reliability and overall effectiveness of two different methods for motivating patients to take aspirin to prevent stroke and heart attacks as well as to develop a plan for translating the intervention into a process that is suitable for a paper-based clinic.

ELIGIBILITY:
Inclusion Criteria:

Patients with an appointment in the Geisinger clinic who:

* are between the ages of 45-70 (male) or 50-70 (female), and
* have one of the following risk factors:

  1. Smoke
  2. Direct LDL > 160 mg/dl
  3. HDL < 45 mg/dl (males) HDL < 35 mg/dl (females)
  4. Diabetes diagnosis
  5. Hypertension diagnosis
  6. CAD diagnosis

Exclusion Criteria:

* > 70 years
* Stomach Ulcer History
* Aspirin Allergy
* Anti-coagulation Therapy History
* Clotting Disorder Diagnosis
* Hypersensitivity to non-steroidal anti-inflammatory agents such as Ibuprofen, Aleve, or Motrin
* Hemorrhagic Stroke History
* Current Aspirin use
* 1st Outpatient Visit

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Aspirin Use At Two Week Follow-Up (Measures Taken at Baseline and Follow-Up) | Two Weeks

SECONDARY OUTCOMES:
Patient Knowledge of Risks/Benefits of Aspirin | Two Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nirav R Shah, MD, MPH, Principal Investigator — Geisinger Clinic
Locations (3):
- United States (3):
  - Geisinger Clinic - Lewistown, Lewistown, Pennsylvania
  - Geisinger Clinic - Moshannon Valley, Philipsburg, Pennsylvania
  - Geisinger Clinic - Lake Scranton, Scranton, Pennsylvania

REFERENCES:
- See also: (Click here for more information about Geisinger Health System) — http://www.geisinger.org